CLINICAL TRIAL: NCT03521700
Title: A Prospective, Randomized Trial to Compare Effects of Intensive Versus Conventional Lipid-lowering Therapy in Patients With Severe Atherosclerotic Renal Artery Stenosis Undergoing Stent Placement
Brief Title: Compare Effects of Intensive Versus Conventional Lipid-lowering Therapy in Patients With Severe Atherosclerotic Renal Artery Stenosis Undergoing Stent Placement
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Xiongjing Jiang, Professor, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-ZX13
Record Dates: First submitted 2018-04-29; First posted 2018-05-11 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Renal Artery Obstruction; Stents; Lipids; Glomerular Filtration Rate; Blood Pressure
Keywords: Renal Artery Obstruction; Stents; Glomerular filtration rate
MeSH Terms: conditions — Renal Artery Obstruction | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: Intensive lipid lowering gourp:10 mg/d rosuvastatin was initially prescribed and target LDL-C was < 1.8mmol/L; Conventional lipid lowering: 5 mg/d rosuvastatin was initially prescribed and target LDL-C was ≥1.8mmol/L, <3.3mmol/L
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive lipid lowering group (Experimental): 10 mg/d rosuvastatin was initially prescribed and target LDL-C was < 1.8mmol/L
  Interventions: Drug: Rosuvastatin
- Conventional lipid lowering group (Other): 5 mg/d rosuvastatin was initially prescribed and target LDL-C was ≥1.8mmol/L, <3.3mmol/L
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — For patients who were assigned to receive intensive lipid lowering, 10 mg/d rosuvastatin was initially prescribed and target LDL-C was < 1.8mmol/L. For patients who were assigned to receive conventional lipid lowering, 5 mg/d rosuvastatin was initially prescribed and target LDL-C was ≥1.8mmol/L, <3.3mmol/L.

SUMMARY:
Although expert consensuses recommend the use of statins in the treatment of atherosclerotic renal artery stenosis, in patients with severe atherosclerotic renal artery stenosis undergoing stent placement, the related investigation focused on renal protection by intensive lipid-lowering therapy is scant , and the optimal target level for lipid reduction remain uncertain. Therefore, we hypothesized that intensive lipid lowering could offer more benefits with respect to renal function in the patients with percutaneous renal artery stenting. We conducted the prospective randomized unblinded trial to compare the renal-protective effect of intensive lipid lowering with that of conventional lipid lowering in patients underwent renal artery stenting (75 patients in each study group)

ELIGIBILITY:
Inclusion Criteria:

1. Angiographic evidence of severe atherosclerotic renal artery stenosis (diameter reduction≥ 70%) with ≥ 20 mmHg systolic translesional gradient or positive captopril renography in the target kidney;
2. Sustained systolic blood pressure ≥ 180 mmHg, and/or diastolic blood pressure ≥ 110 mmHg while not receiving drug therapy or systolic blood pressure ≥ 140 mmHg, and/or diastolic blood pressure ≥ 90mmHg while taking standard triple-drug combination treatment (including one diuretic);
3. Estimated glomerular filtration rate≥ 10 ml/min/1.73m2 with longitudinal kidney length ≥ 7 cm supplied by target artery;
4. Serum creatinine level<264umol/L；
5. Urine protein≤ 1+

Exclusion Criteria:

1. Allergy to rosuvastatin;
2. Myopathy;
3. Active liver disease or alanine aminotransferase and/or aspartate aminotransferase levels ≥ three times the upper limit of normality;
4. Serious perioperative complications;
5. Severe chronic congestive heart failure (New York Heart Association functional class IV );
6. Patients who should be excluded basing on physician discretion.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2014-12-30 (Actual); Study Completion 2015-12-30 (Actual)

PRIMARY OUTCOMES:
Change in estimated glomerular filtration rate | 12 months after randomization

SECONDARY OUTCOMES:
Change in urinary albumin-creatinine ratio | 12 months after randomization
Change in the number of antihypertensive medications | 12 months after randomization
Change in systolic blood pressure | 12 months after randomization
Change in diastolic blood pressure | 12 months after randomization
Stent restenosis rate | 12 months after randomization
Major clinical events | 12 months after randomization
  death from cardiovascular or renal causes, myocardial infarction, hospitalization for congestive heart failure, stroke, and a relative increase in SCr from baseline of ≥50%

CONTACTS AND LOCATIONS:
Overall Officials: Xiongjing Jiang, MD, Principal Investigator — Fuwai Hospital, National Center for Cardiovascular Disease, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Fuwai Hospital, National Center for Cardiovascular Disease, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China